CLINICAL TRIAL: NCT02668770
Title: A Phase I Trial of Ipilimumab (Immunotherapy) and MGN1703 (TLR Agonist) in Patients With Advanced Solid Malignancies
Brief Title: Ipilimumab (Immunotherapy) and MGN1703 (TLR Agonist) in Patients With Advanced Solid Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Mologen AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0135; NCI-2016-00276 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Advanced Cancers; Melanoma
Keywords: Advanced Cancers; Melanoma; Advanced solid malignancies; Metastatic; MGN1703; Ipilimumab; Yervoy; BMS-734016; MDX010; Refractory; Relapsed
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Recurrence | interventions — MGN1703; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation Group: MGN1703 + Ipilimumab (Experimental): Participants receive MGN1703 on Days 1, 8, and 15 of all cycles as an injection under the skin. Ipilimumab dosed at 3 mg/kg once per cycle on Day 8 following MGN1703 administration.
  Each cycle is 21 days long. Participants receive a total of 4 treatment cycles for a total of 12 weeks on treatment.
  Interventions: Drug: MGN1703; Drug: Ipilimumab
- MTD Group: MGN1703 (subcutaneously) + Ipilimumab (Experimental): Dose expansion group consists of participants with advanced malignancy and cutaneous or subcutaneous manifestations.
  MGN1703 given subcutaneously at MTD from the Dose Escalation Group. Ipilimumab dosed at 3 mg/kg once per cycle on Day 8 following MGN1703 administration.
  Each cycle is 21 days long.
  Interventions: Drug: MGN1703; Drug: Ipilimumab
- MTD Group: MGN1703 (intratumoral injection) + Ipilimumab (Experimental): Dose expansion group consists of participants with advanced malignancy and cutaneous or or subcutaneous manifestations.
  MGN1703 given by intratumoral injection at MTD from the Dose Escalation Group. Ipilimumab dosed at 3 mg/kg once per cycle on Day 8 following MGN1703 administration.
  Each cycle is 21 days long.
  Interventions: Drug: MGN1703; Drug: Ipilimumab
- MTD Post XRT Group: MGN1703 (subcutaneously) + Ipilimumab (Experimental): Dose expansion group consists of participants with advanced malignancy treated with radiation (XRT) within the past 2 weeks.
  MGN1703 given subcutaneously at MTD from the Dose Escalation Group. Ipilimumab dosed at 3 mg/kg once per cycle on Day 8 following MGN1703 administration.
  Each cycle is 21 days long.
  Interventions: Drug: MGN1703; Drug: Ipilimumab

INTERVENTIONS:
Drug: MGN1703 — Dose Escalation Group Starting Dose: 15 mg on Days 1, 8, and 15 of each 21 day cycle.
  Dose Expansion Group Starting Dose: Maximum tolerated dose from Dose Escalation Group.
Drug: Ipilimumab — Dose Escalation and Dose Expansion Group Dose: 3 mg/kg by vein on Day 8 of a 21 day cycle.
  Other Names: BMS-734016; Yervoy; MDX010

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of MGN1703 that can be given in combination with ipilimumab to patients with advanced tumors. The safety of this drug combination will also be studied.

This is an investigational study. MGN1703 is not FDA approved or commercially available. It is currently being used for research purposes only. Ipilimumab is FDA approved and commercially available for the treatment of unresectable (cannot be removed with surgery) or metastatic (has spread) melanoma.

Up to 60 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of MGN1703 based on when you joined this study. Up to 4 dose levels of MGN1703 will be tested. Up to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level of MGN1703. Each new group will receive a higher dose of MGN1703 than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of MGN1703 is found. This is called dose escalation.

In another part of the study (called dose expansion) up to 3 groups of up to 12 additional participants will be enrolled. Two (2) groups will receive MGN1703 at the highest tolerable dose that was found in dose escalation. One (1) group will receive the first dose level of MGN1703 (if it is found to be tolerable). The study doctor will tell you which dose of MGN1703 you will receive.

All participants will receive the same dose level of ipilimumab. You will receive ipilimumab at standard doses.

Study Drug Administration:

Each study cycle is 21 days.

You will be given MGN1703 as an injection under the skin on Days 1, 8, and 15 of each cycle. Each administration will be between 1-4 injections in multiple parts of your body (such as your upper arms and thighs, your abdomen and thighs, or your abdomen and upper arms). The study doctor will tell you how many times you will be injected.

If you are in dose expansion, you may receive MGN1703 as an injection directly into the tumor. The study doctor will tell you if you will receive the study drug this way.

You will also receive ipilimumab by vein over about 90 minutes on Day 8 of Cycles 1-4.

Study Visits:

During Week 1 of every cycle, blood (about 1 teaspoon) will be drawn for routine tests.

During Week 2 of Cycles 1-4, you will have a physical exam.

During Week 3 of Cycles 1 and 3, blood (about 5 teaspoons) will be drawn for routine tests and biomarker testing.

During Week 3 of Cycles 2 and 4:

* Blood (about 5 teaspoons) will be drawn for routine tests and biomarker testing.
* Urine will be collected for routine tests.
* You will have an EKG.
* You will have imaging scans to check the status of the disease.
* If you can become pregnant, blood (about 1 teaspoon) will be drawn for a pregnancy test.

If you are in dose expansion and depending on when you join the study, on Day 1 of Cycle 3 you will have a biopsy for biomarker testing (including genetic biomarkers).

During Cycle 4 and then every even-numbered cycle after that (Cycles 6, 8, 10, and so on):

* You will have a physical exam.
* Blood (about 5 teaspoons) will be drawn for routine tests and biomarker testing.
* You will have imaging scans to check the status of the disease. After 1 year on study, you will have these scans every 4 cycles.

During Cycle 4 and then every 4 cycles after that (Cycles 8, 12, 16, and so on):

* Urine will be collected for routine tests.
* You will have an EKG.
* If you can become pregnant, blood (about 1 teaspoon) will be drawn for a pregnancy test.

Every 30 days for 90 days after your last dose of study drug, you will be called by a member of the study staff and asked about any new anticancer drugs you may have started and how you are feeling. You may also be asked these questions during a routine clinic visit or this information may be collected from your medical record. If you are called, each call should last about 10-15 minutes.

Length of Study:

You may receive MGN1703 in combination with ipilimumab for up to 4 cycles. After that, you may continue taking MGN1703 alone for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

You participation on this study will be over 90 days after your last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically-confirmed metastatic or locally advanced solid tumor that has failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist.
2. There is no limit on the number of prior treatment regimens.
3. Patients must be off prior chemotherapy, hormonal therapy, or biological therapy for at least 4 weeks or >3 half-lives whichever comes first. Patients with prostate cancer may continue to receive LHRH agonist (unless orchiectomy has been performed).
4. ECOG performance status </= 2 (Karnofsky >60%).
5. Patients must have adequate organ and marrow function as defined below within 7 days: WBC >/= 2500/mm^3. Absolute neutrophil count (ANC) >/= 1,500/mm^3. Absolute lymphocyte count (ALC) >/= 500/mm^3. Hemoglobin >/= 9g/dl. Platelets >/= 75,000/mm^3. Creatinine </= 2.0 x ULN or measured CrCl of >/= 50ml/m^2/1.73 m^2. Total bilirubin </= 2.0 mg/dL (unless previously diagnosed with Gilbert's Syndrome). AST(SGOT)/ALT(SGPT) </= 3 times the institutional upper limit of normal (patients with liver involvement will be allowed </= 5.0 X institutional upper normal limit).
6. Patients must have recovered from toxicity related to prior therapy to at least grade 1 (defined by CTCAE 4.0) or baseline level. Chronic stable grade 2 peripheral neuropathy secondary to neurotoxicity from prior therapies may be considered on a case by case basis by the Principal Investigator.
7. As the effect of these drugs on the developing human fetus is not known, women of child-bearing potential and men must agree to use adequate contraception (abstinence; hormonal or barrier method of birth control) for the study and at least 2 months after completion.
8. Female patient of childbearing potential has a negative serum pregnancy test within 7 days of study enrollment.
9. Patients must be willing and able to review, understand, and provide written consent before study enrollment.
10. Measurable disease as defined by irRC or RECIST 1.1 criteria
11. Age >/= 18 years.

Exclusion Criteria:

1. Severe autoimmune disease: Patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus or autoimmune vasculitis [e.g., Wegener's Granulomatosis] are excluded from this study. Patients with history of mild autoimmune disorders - including but not limited to mild psoriasis or Hashimoto's hyperthyroidism may be included at the discretion of the principle investigator.
2. History of acute diverticulitis, intra-abdominal abscess, GI obstruction, abdominal carcinomatosis or other known risk factors for bowel perforation.
3. Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of AEs: e.g. a condition associated with frequent diarrhea or chronic skin conditions, recent surgery or colonic biopsy from which the patient has not recovered, or partial endocrine organ deficiencies.
4. Current evidence of active and uncontrolled infection, NYHA Class III-IV CHF, documented Child's class B-C cirrhosis, active pancreatitis or uncontrolled medical disease which in the opinion of the investigator could compromise assessment of efficacy.
5. Known human immunodeficiency virus (HIV)-positive and on highly active antiretroviral therapy (HAART), and/or Hepatitis B or C on treatment. Drug interactions between those agents and these experimental agents are wholly unknown (screening not required).
6. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days of day 1 of therapy.
7. Known hypersensitivity to the components of study drugs, its analogs, or drugs of similar chemical or biologic composition.
8. Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to one month prior to or after any dose of ipilimumab).
9. Concomitant therapy with any of the following: IL-2, interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigational therapies; or chronic use of systemic corticosteroids (when used in the management of cancers other than intracranial glioblastoma, gliosarcoma or anaplastic astrocytoma, or when used to treat non-cancer-related illnesses).
10. Radiation therapy within 4 weeks of study enrollment (exception is radiotherapy expansion arm which requires radiation treatment within 2 week period).
11. Pregnant and breastfeeding women are excluded from this study. Women of child-bearing potential and men must agree to use contraception prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician.
12. Use of any other concurrent investigational agents or anticancer agents including hormonal therapy, except in the case of prostate cancer patients who are being treated with LHRH agonist at the time of trial entry.
13. Previous exposure to TLR agonist therapy.
14. Known history of plasma cortisol and adrenocorticotropic hormone (ACTH) levels consistent with adrenal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of MGN1703 with Ipilimumab | 84 days
  If more than or equal to one third of the participants at a dose level experience dose limiting toxicity (DLT), the MTD reassessed and the next lowest dose level for the combination therapy considered the MTD.

SECONDARY OUTCOMES:
Tumor Response | 84 days
  Tumor response defined as one or other of the following: (1) stable disease for more than than or equal to 4 months, (2) decrease in measurable tumor (sentinel lesions) by more than or equal to 20% by irRC criteria.

CONTACTS AND LOCATIONS:
Overall Officials: David S. Hong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Nardo M, Gouda MA, Reilley MJ, Biter AB, Lim J, Bean SA, Nguyen LM, Bhosale PR, Ager CR, Couillault CA, Piha-Paul SA, Fu S, Tsimberidou AM, Yap TA, Naing A, Rodon J, Subbiah V, Karp DD, Curran MA, Hong DS. Lefitolimod in Combination with Ipilimumab in Patients with Advanced Solid Tumors: A Phase I Trial. J Immunother Precis Oncol. 2025 Feb 7;8(2):89-98. doi: 10.36401/JIPO-24-17. eCollection 2025 May. PMID 39959251
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org